CLINICAL TRIAL: NCT02824913
Title: Randomized, Crossover Study of the Pharmacodynamic Activity of P-321 Ophthalmic Solution Compared to Placebo in Subjects With Dry Eye Disease Characterized by Low Tear Volume
Brief Title: Study of the Pharmacodynamic Activity of P-321 Ophthalmic Solution Compared to Placebo in Subjects With Dry Eye Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Parion Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: P-321-201
Record Dates: First submitted 2016-07-01; First posted 2016-07-07 (Estimated); Results first posted 2018-01-19 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2017-12

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- P-321 Ophthalmic Solution (Experimental): 0.017% P-321 Ophthalmic Solution will be administered to approximately 8 patients in Phase I and either 0.05% P-321 Ophthalmic Solution or 0.01% P-321 Ophthalmic Solution or additional 0.017% P-321 Ophthalmic Solution will be administered to approximately 16 patients in Phase II
  Interventions: Drug: P-321 Ophthalmic Solution
- Drug: P-321 Ophthalmic Solution placebo (Placebo Comparator): Placebo treatment administered to approximately 8 patients in Phase I and approximately 16 patients in Phase II
  Interventions: Drug: P-321 Ophthalmic Solution placebo

INTERVENTIONS:
Drug: P-321 Ophthalmic Solution
  Other Names: P-321
  Arms: P-321 Ophthalmic Solution
Drug: P-321 Ophthalmic Solution placebo
  Other Names: Placebo Comparator; Placebo
  Arms: Drug: P-321 Ophthalmic Solution placebo

SUMMARY:
The purpose of this Phase 2a study is to assess changes in tear volume by the non-invasive techniques Ultra High Resolution Optical Coherence Tomography (UHR-OCT) following the administration of P-321 Ophthalmic Solution or Placebo in subjects with tear deficient dry eye disease.

DETAILED DESCRIPTION:
This is a single-center, randomized, cross-over placebo controlled study to evaluate the changes in tear volume by P-321 Ophthalmic Solution and Placebo. The study will enroll subjects with tear deficient dry eye disease to receive sequentially one of two treatment sequences: P-321 Ophthalmic Solution then Placebo or Placebo then P-321. The study will consist of two Phases: In each Phase, subjects will be treated with P-321 Ophthalmic Solution under the same study design.

Approximately twenty-four eligible subjects will complete the study with approximately 8 subjects participating in Phase 1 and the remainder of the 24 subjects participating in the phase 2. Decisions on the dose to be used in Phase 2 will be made based on Phase 1 data.

The study will consist of three study visits: a Screening Visit (Visit 1), and two treatment visits (Visit 2 and Visit 3). The primary and secondary outcome measures will be assessed at each treatment visit. Safety assessments include adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Male or female subjects aged 18 to 80 years
3. Have a history of predominantly tear-deficient dry eye of mild to moderate severity, supported by a previous clinical diagnosis
4. Have normal lid anatomy
5. Subjects must:

   1. Remain on current medications for the duration of the study and have been on the current medication regimen at least during the past 28 days

Exclusion Criteria:

1. Have undergone refractive eye surgery in either eye during the past 12 months
2. Have undergone uncomplicated cataract surgery in either eye during the past 3 months
3. Have undergone previous eyelid surgery in either eye (External blepharoplasty, not resulting in exposure or abnormal blinking is allowed)
4. Have undergone botulinum toxin (BotoxTh1 or equivalent) injection in the periocular area within 3 months prior to Visit 1
5. Subjects that have a systemic, multi-organ disease requiring active medical or surgical treatment are excluded with the exception of subjects with SS or GVHD
6. Have punctal plugs, punctal occlusion, history of nasolacrimal duct obstruction or wear scleral lens.
7. Past or present exposure keratopathy, neurotrophic keratopathy, lagophthalmos, or trichiasis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Boyer, Study Director — Parion Sciences
Locations (1):
- Bascom Palmer Eye Institute, University of Miami Health System, Plantation, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- P-321 Ophthalmic Solution Then Placebo Comparator: At Visit 2 0.017% P-321 Ophthalmic Solution will be administered to approximately 8 patients in Phase I and either 0.05% P-321 Ophthalmic Solution or 0.01% P-321 Ophthalmic Solution or additional 0.017% P-321 Ophthalmic Solution will be administered to approximately 16 patients in Phase II
  After a washout period of 7-14 days at Visit 3 Placebo Comparator will be administered to approximately 8 patients in Phase I and approximately 16 patients in Phase II
- Placebo Comparator Then P-321 Ophthalmic Solution: At Visit 2 Placebo treatment will be administered to approximately 8 patients in Phase I and approximately 16 patients in Phase II
  After a washout period of 7-14 days at Visit 3 0.017% P-321 Ophthalmic Solution will be administered to approximately 8 patients in Phase I and either 0.05% P-321 Ophthalmic Solution or 0.01% P-321 Ophthalmic Solution or additional 0.017% P-321 Ophthalmic Solution will be administered to approximately 16 patients in Phase II
Period: First Intervention (1 Day)
Arm/Group | P-321 Ophthalmic Solution Then Placebo Comparator | Placebo Comparator Then P-321 Ophthalmic Solution
Started | 1 | 0
Completed | 1 (Only one subject was enrolled in the study and received both study treatments.) | 0
Not Completed | 0 | 0
Period: Washout (7-14 Days)
Arm/Group | P-321 Ophthalmic Solution Then Placebo Comparator | Placebo Comparator Then P-321 Ophthalmic Solution
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | P-321 Ophthalmic Solution Then Placebo Comparator | Placebo Comparator Then P-321 Ophthalmic Solution
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only one patient was enrolled in the study, the patient was randomized into the Group of P-321 Ophthalmic Solution Then Placebo Comparator. No patients participated in the Group of Placebo Comparator Then P-321 Ophthalmic Solution
Groups:
- P-321 Ophthalmic Solution Then Placebo Comparator: At Visit 2 0.017% P-321 Ophthalmic Solution will be administered to approximately 8 patients in Phase I and either 0.05% P-321 Ophthalmic Solution or 0.01% P-321 Ophthalmic Solution or additional 0.017% P-321 Ophthalmic Solution will be administered to approximately 16 patients in Phase II P-321 Ophthalmic Solution
  At Visit 3 Placebo comparator will be administered to approximately 8 patients in Phase I and approximately 16 patients in Phase II
- Placebo Comparator Then P-321 Ophthalmic Solution: At Visit 2 Placebo comparator will be administered to approximately 8 patients in Phase I and approximately 16 patients in Phase II
  At Visit 3 0.017% P-321 Ophthalmic Solution will be administered to approximately 8 patients in Phase I and either 0.05% P-321 Ophthalmic Solution or 0.01% P-321 Ophthalmic Solution or additional 0.017% P-321 Ophthalmic Solution will be administered to approximately 16 patients in Phase II P-321 Ophthalmic Solution
- Total: Total of all reporting groups
Arm/Group | P-321 Ophthalmic Solution Then Placebo Comparator | Placebo Comparator Then P-321 Ophthalmic Solution | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Tear Meniscus Volume Following the Administration of P-321 Ophthalmic Solution or Placebo
Description: Tear meniscus volume, from measurements of tear meniscus area by UHR-OCT and the length of the eyelid was estimated over time (0 to 6 hours) following administration of placebo or P-321 Ophthalmic Solution.
Time Frame: Pre-dose and up to six hours after dose
Population: One subject enrolled in the study. Subject received both study treatments (a single instillation of 0.017% P-321 Ophthalmic Solution in both eyes and a single instillation of Placebo in both eyes).
  Study was terminated, raw data obtained. Processing of data was not conducted to obtain primary and secondary outcomes, therefore none reported.
Arm/Group | P-321 Ophthalmic Solution Then Placebo Comparator | Placebo Comparator Then P-321 Ophthalmic Solution
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Lower Tear Meniscus Height as Measured by the Keratograph 5M
Description: Tear meniscus height of the inferior eyelid was measured with the Keratograph 5M over time (0 to 6 hours) following the administration of placebo or P-321 Ophthalmic Solution
Time Frame: Pre-dose and up to six hours after dose
Population: as for outcome 1
Arm/Group | P-321 Ophthalmic Solution Then Placebo Comparator | Placebo Comparator Then P-321 Ophthalmic Solution
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Comparison of Lower Tear Meniscus Height Measurements Between UHR-OCT and Keratograph 5M
Description: Tear meniscus height of the inferior eyelid was measured by UHR-OCT and Keratograph 5M over time (0 to 6 hours) following the administration of placebo or P-321 Ophthalmic Solution
Time Frame: Pre-dose and up to six hours after dose
Population: as for outcome 1
Arm/Group | P-321 Ophthalmic Solution Then Placebo Comparator | Placebo Comparator Then P-321 Ophthalmic Solution
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Adverse Events
Description: Number of patients experiencing adverse events comparing P-321 to placebo
Time Frame: 2 or 7 hours
Population: One subject enrolled in the study. Subject received both study treatments (a single instillation of 0.017% P-321 Ophthalmic Solution in both eyes and a single instillation of Placebo in both eyes).
Measure: Count of Participants; unit: Participants
Arm/Group | P-321 Ophthalmic Solution Then Placebo Comparator | Placebo Comparator Then P-321 Ophthalmic Solution
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Subjects were to receive 2 treatments (P-321 Ophthalmic Solution and Placebo) during this study; first treatment on Visit 2 (3 to 9 days after screening) and second treatment on Visit 3 (7 to 14 days after the first treatment).
Description: An AE was defined as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product, which did not necessarily have to have a causal relationship with this treatment. A treatment-emergent AE (TEAE) was an AE that either commenced following initiation of study treatment or was present prior to study treatment but increased in frequency or severity following initiation of study treatment.
Groups:
- P-321 Ophthalmic Solution: 0.017% P-321 Ophthalmic Solution will be administered to approximately 8 patients in Phase I and either 0.05% P-321 Ophthalmic Solution or 0.01% P-321 Ophthalmic Solution or additional 0.017% P-321 Ophthalmic Solution will be administered to approximately 16 patients in Phase II
  P-321 Ophthalmic Solution
- Drug: P-321 Ophthalmic Solution Placebo: Placebo treatment administered to approximately 8 patients in Phase I and approximately 16 patients in Phase II
  P-321 Ophthalmic Solution placebo
Arm/Group | P-321 Ophthalmic Solution | Drug: P-321 Ophthalmic Solution Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator may publish or present the results based on data generated at their Institution, provided that: (a) Sponsor publishes the results from all sites participating in the Study; (b) Institution receives notification from Sponsor that publication of the multi-site results is no longer planned; or (c) twelve (12) months following the close of study, whichever occurs first.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT02824913/Prot_SAP_000.pdf